CLINICAL TRIAL: NCT02911831
Title: IV Tranexamic Acid Prior to Hysterectomy for Reduction of Intraoperative Blood Loss: A Randomized Placebo-Controlled Trial
Brief Title: IV Tranexamic Acid Prior to Hysterectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Magdy Milad, MD, Chief of Minimally Invasive Gynecologic Surgery in the Department of Obstetrics and Gynecology Albert B. Gerbie, MD, Professor of Obstetrics and Gynecology Professor of Obstetrics and Gynecology (Minimally Invasive Gynecologic Surgery), Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU00203110
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2021-09

CONDITIONS: Hysterectomy; Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid: Abdominal Hysterectomy (Experimental): Agent/Device: Tranexamic acid. Patients undergoing abdominal hysterectomy who consent to the study may be randomized to this arm.
  · Protocol dose: 1g in solution to be given intravenously, within 1 hour prior to procedure
  Interventions: Drug: Tranexamic Acid
- Sodium chloride (placebo): Abdominal Hysterectomy (Placebo Comparator): Agent/Device: 0.9% sodium chloride solution. Patients undergoing abdominal hysterectomy who consent to the study may be randomized to this arm.
  · Protocol dose: 100ml to be given intravenously, within 1 hour prior to procedure
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: Tranexamic Acid
  Other Names: TXA
  Arms: Tranexamic Acid: Abdominal Hysterectomy
Drug: Sodium Chloride
  Other Names: Normal saline
  Arms: Sodium chloride (placebo): Abdominal Hysterectomy

SUMMARY:
The objective of this study is to determine the effect of 1g of IV tranexamic acid given within 1 hour pre-operatively on intraoperative blood loss at time of hysterectomy.

DETAILED DESCRIPTION:
Tranexamic acid (TXA) is a synthetic lysine analog that inhibits plasmin fibrinolysis. It may be administered orally, intravenously, or topically, with a rapid onset of action (tmax = appx 3 hours) and 11-hour half-life. It is 6 to 10 times more potent than aminocaproic acid, another commonly used synthetic antifibrinolytic agent. Typical IV dosing is 10 mg/kg followed by infusion of 1mg/kg/hour, or simply 1g intravenously in one dose.

The efficacy of tranexamic acid in control of hemorrhage in trauma patients has been reported extensively. The CRASH-2 trial collaborators randomized 20,211 adult trauma patients with significant bleeding or at risk of significant bleeding within 8 hours of injury to IV tranexamic acid or placebo. All-cause mortality was significantly reduced with tranexamic acid (RR .91; p = .0035). Additionally, risk of death due to bleeding was significantly lower in those receiving tranexamic acid (RR .85; p = .0077). No differences in risk of vascular occlusive events were noted. Further analysis revealed reduced risk of death from bleeding if TXA was given within 3 hours of injury; treatment administered after 3 hours from injury increased the risk of death due to bleeding.

Administration of TXA during elective surgery has also been investigated. A 2011 systematic review of 252 randomized trials of patients undergoing elective surgery across disciplines included administration of TXA, aminocaproic acid, and aprotinin. TXA administration reduced the risk of transfusion peri-operatively (RR .61). A 2012 meta-analysis of TXA use in both elective an emergency surgery revealed that TXA reduced the risk of transfusion by one-third. The effect of TXA on risk of myocardial infarction, deep vein thrombosis, and pulmonary embolism was not statistically significant.

The utility of TXA appears to extend to obstetric hemorrhage. Several published studies exist analyzing its use in prevention of postpartum hemorrhage, though the drug is not considered standard for prevention or treatment of this condition. A pilot randomized open-label trial of IV TXA in women with postpartum hemorrhage over 800cc reported a lower median blood loss between groups, though the effect was modest. Additionally, significantly fewer women in the TXA group required transfusion or invasive procedures. A recent Cochrane review reports on twelve trials of low risk women undergoing cesarean section or spontaneous birth who received uterotonics with or without the addition of TXA. TXA was effective in decreasing estimated blood loss over 1 liter in women undergoing cesarean section. Mean blood loss was significantly lower in women receiving TXA (mean difference -77.79mL); effect was similar for women undergoing cesarean section and vaginal birth. Finally, the WOMAN trial is a large, ongoing, placebo-controlled trial examining the effect of early TXA administration in clinically diagnosed postpartum hemorrhage.

The use of TXA in the management of acute and abnormal uterine bleeding has been reported, and is FDA-approved for treatment of menorrhagia. One randomized study of oral TXA in the treatment of ovulatory menorrhagia reported a 45% decrease in mean menstrual blood loss with use of TXA as compared with placebo. Other studies have echoed these findings, with TXA more effective than NSAIDs but less effective than the levonorgestrel intrauterine device (IUD) in decreasing menstrual blood loss. More recently, a double-blind, placebo-controlled randomized-controlled trial (RCT) confirmed a significant decrease in menstrual blood loss(mean -69cc), improvements in social/physical limitations caused by menorrhagia and self-perceived menstrual blood loss. No data exist examining the efficacy of IV TXA in the management of acute or severe uterine bleeding.

Few studies have specifically examined the utility of prophylactic TXA in reducing mean blood loss during hysterectomy or other gynecologic procedures. In one study of patients undergoing endometrial ablation and endoscopic endometrial resection, intraoperative and postoperative IV TXA significantly decreased total blood loss. In patients undergoing major debulking surgery for gynecologic cancers, administration of IV TXA has been shown to decrease intra-operative blood loss by 30%. One well-designed study of women with advanced-stage ovarian cancer randomized patients to 15 mg/kg IV TXA or the same volume of placebo immediately before surgery. Outcomes included significantly lower mean estimated blood loss and decreased need for transfusion in the TXA group.

This study sought to determine whether a single preoperative dose of IV tranexamic acid effectively reduces intraoperative blood loss and need for transfusion in patients undergoing laparoscopic, abdominal, or vaginal hysterectomy for benign indications.

Objective:

To determine the effect of 1g of IV tranexamic acid given within 1 hour pre-operatively on intraoperative blood loss at time of hysterectomy.

Primary endpoint:

Estimated blood loss as determined by anesthesia and surgeon at time of hysterectomy, difference between post-operative and pre-operative hemoglobin, length of hospital stay, length of procedure, need for blood transfusion and post-operative venous thromboembolic events.

Treatment Dosage and Administration:

1g IV tranexamic acid or 100ml 0.9% sodium chloride solution administered within 1 hour of the start of the procedure

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting for hysterectomy for any benign indication including but not limited to abnormal uterine bleeding, menorrhagia, uterine fibroids, adenomyosis, pelvic pain, dysmenorrhea, pelvic organ prolapse or endometriosis.
2. Age ≥ 18 years
3. Pre-operative hemoglobin >8 g/dl
4. Willing to have IV tranexamic acid or a placebo prior to hysterectomy
5. Ability to understand and the willingness to sign a written informed consent.
6. Can be previously treated with Depo-Lupron, Depo-Provera, Oral Contraceptive pills, Mirena IUD, endometrial ablation, myomectomy, oral progestins
7. Hysterectomy in combination with the following procedures is permitted: unilateral/bilateral salpingectomy or oophorectomy, ovarian cystectomy, fulguration/excision of endometriosis, appendectomy, sacrocolpopexy, anterior/posterior repair, uterosacral vault suspension, retropubic midurethral sling and cystoscopy

Exclusion Criteria:

1. Patients with known or suspected endometrial/ovarian/cervical cancer.
2. Patients undergoing hysterectomy for endometrial hyperplasia or cervical dysplasia.
3. Patients currently undergoing treatment for any type of cancer.
4. Patients with known bleeding/clotting disorders or a history of thromboembolism (including deep venous thrombosis or pulmonary embolism)
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to tranexamic acid.
6. Any procedures which occur in combination with other elective surgical procedures (such as abdominoplasty, breast augmentation, etc) which are not included in the previously mentioned inclusion criteria above will be excluded from data analysis.
7. Uncontrolled current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, subarachnoid hemorrhage, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Patients with acquired defective color vision
9. Patients with known renal failure and/or Cr > 5 within the last 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Intra-operative blood loss | Intra-operative

SECONDARY OUTCOMES:
Change in hemoglobin, postoperative from baseline | < 12 hours
Need for blood transfusion | Intra-operative
Length of hospital stay | <1 week
Length of operative procedure | <12 hours
Rates of postoperative thromboembolic events | 12 weeks
Incidence of drug-related adverse events | 12 weeks
Health care cost | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Milad, MD, Principal Investigator — Northwestern University, Northwestern Memorial Hopsital
Locations (1):
- Northwestern University - Northwestern Medicine, Lavin Family Pavillion, Chicago, Illinois, United States

REFERENCES:
- [Background] Walsh CA, Walsh SR, Tang TY, Slack M. Total abdominal hysterectomy versus total laparoscopic hysterectomy for benign disease: a meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2009 May;144(1):3-7. doi: 10.1016/j.ejogrb.2009.01.003. Epub 2009 Mar 25. PMID 19324491
- [Background] Nieboer TE, Johnson N, Lethaby A, Tavender E, Curr E, Garry R, van Voorst S, Mol BW, Kluivers KB. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD003677. doi: 10.1002/14651858.CD003677.pub4. PMID 19588344
- [Background] Taggart DP, Siddiqui A, Wheatley DJ. Low-dose preoperative aspirin therapy, postoperative blood loss, and transfusion requirements. Ann Thorac Surg. 1990 Sep;50(3):424-8. doi: 10.1016/0003-4975(90)90488-r. PMID 2400264
- [Background] Carson JL, Duff A, Poses RM, Berlin JA, Spence RK, Trout R, Noveck H, Strom BL. Effect of anaemia and cardiovascular disease on surgical mortality and morbidity. Lancet. 1996 Oct 19;348(9034):1055-60. doi: 10.1016/S0140-6736(96)04330-9. PMID 8874456
- [Background] Okuyama M, Ikeda K, Shibata T, Tsukahara Y, Kitada M, Shimano T. Preoperative iron supplementation and intraoperative transfusion during colorectal cancer surgery. Surg Today. 2005;35(1):36-40. doi: 10.1007/s00595-004-2888-0. PMID 15622462
- [Background] Sesti F, Ticconi C, Bonifacio S, Piccione E. Preoperative administration of recombinant human erythropoietin in patients undergoing gynecologic surgery. Gynecol Obstet Invest. 2002;54(1):1-5. doi: 10.1159/000064688. PMID 12297709
- [Background] Lethaby A, Vollenhoven B, Sowter M. Pre-operative GnRH analogue therapy before hysterectomy or myomectomy for uterine fibroids. Cochrane Database Syst Rev. 2001;(2):CD000547. doi: 10.1002/14651858.CD000547. PMID 11405968
- [Background] Okamoto S, Okamoto U. Amino-methyl-cyclohexane-carboxylic acid: AMCHA: a new potent inhibitor of fibrinolysis. Keio J Med. 1962;11:105-115.
- [Background] Roberts I, Prieto-Merino D. Applying results from clinical trials: tranexamic acid in trauma patients. J Intensive Care. 2014 Oct 5;2(1):56. doi: 10.1186/s40560-014-0056-1. eCollection 2014. PMID 25705414
- [Background] Dunn CJ, Goa KL. Tranexamic acid: a review of its use in surgery and other indications. Drugs. 1999 Jun;57(6):1005-32. doi: 10.2165/00003495-199957060-00017. PMID 10400410
- [Background] Sundstrom A, Seaman H, Kieler H, Alfredsson L. The risk of venous thromboembolism associated with the use of tranexamic acid and other drugs used to treat menorrhagia: a case-control study using the General Practice Research Database. BJOG. 2009 Jan;116(1):91-7. doi: 10.1111/j.1471-0528.2008.01926.x. Epub 2008 Nov 11. PMID 19016686
- [Background] Berntorp E, Follrud C, Lethagen S. No increased risk of venous thrombosis in women taking tranexamic acid. Thromb Haemost. 2001 Aug;86(2):714-5. No abstract available. PMID 11522029
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] CRASH-2 collaborators; Roberts I, Shakur H, Afolabi A, Brohi K, Coats T, Dewan Y, Gando S, Guyatt G, Hunt BJ, Morales C, Perel P, Prieto-Merino D, Woolley T. The importance of early treatment with tranexamic acid in bleeding trauma patients: an exploratory analysis of the CRASH-2 randomised controlled trial. Lancet. 2011 Mar 26;377(9771):1096-101, 1101.e1-2. doi: 10.1016/S0140-6736(11)60278-X. PMID 21439633
- [Background] Henry DA, Carless PA, Moxey AJ, O'Connell D, Stokes BJ, Fergusson DA, Ker K. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2011 Mar 16;2011(3):CD001886. doi: 10.1002/14651858.CD001886.pub4. PMID 21412876
- [Background] Ker K, Edwards P, Perel P, Shakur H, Roberts I. Effect of tranexamic acid on surgical bleeding: systematic review and cumulative meta-analysis. BMJ. 2012 May 17;344:e3054. doi: 10.1136/bmj.e3054. PMID 22611164
- [Background] Ducloy-Bouthors AS, Jude B, Duhamel A, Broisin F, Huissoud C, Keita-Meyer H, Mandelbrot L, Tillouche N, Fontaine S, Le Goueff F, Depret-Mosser S, Vallet B; EXADELI Study Group; Susen S. High-dose tranexamic acid reduces blood loss in postpartum haemorrhage. Crit Care. 2011;15(2):R117. doi: 10.1186/cc10143. Epub 2011 Apr 15. PMID 21496253
- [Background] Novikova N, Hofmeyr GJ, Cluver C. Tranexamic acid for preventing postpartum haemorrhage. Cochrane Database Syst Rev. 2015 Jun 16;2015(6):CD007872. doi: 10.1002/14651858.CD007872.pub3. PMID 26079202
- [Background] Shakur H, Elbourne D, Gulmezoglu M, Alfirevic Z, Ronsmans C, Allen E, Roberts I. The WOMAN Trial (World Maternal Antifibrinolytic Trial): tranexamic acid for the treatment of postpartum haemorrhage: an international randomised, double blind placebo controlled trial. Trials. 2010 Apr 16;11:40. doi: 10.1186/1745-6215-11-40. PMID 20398351
- [Background] Preston JT, Cameron IT, Adams EJ, Smith SK. Comparative study of tranexamic acid and norethisterone in the treatment of ovulatory menorrhagia. Br J Obstet Gynaecol. 1995 May;102(5):401-6. doi: 10.1111/j.1471-0528.1995.tb11293.x. PMID 7612535
- [Background] Milsom I, Andersson K, Andersch B, Rybo G. A comparison of flurbiprofen, tranexamic acid, and a levonorgestrel-releasing intrauterine contraceptive device in the treatment of idiopathic menorrhagia. Am J Obstet Gynecol. 1991 Mar;164(3):879-83. doi: 10.1016/s0002-9378(11)90533-x. PMID 1900665
- [Background] Lukes AS, Moore KA, Muse KN, Gersten JK, Hecht BR, Edlund M, Richter HE, Eder SE, Attia GR, Patrick DL, Rubin A, Shangold GA. Tranexamic acid treatment for heavy menstrual bleeding: a randomized controlled trial. Obstet Gynecol. 2010 Oct;116(4):865-875. doi: 10.1097/AOG.0b013e3181f20177. PMID 20859150
- [Background] Ergun B, Bastu E, Ozsurmeli M, Celik C. Tranexamic acid: a potential adjunct to resectoscopic endometrial ablation. Int Surg. 2012 Oct-Dec;97(4):310-4. doi: 10.9738/CC149.1. PMID 23294071
- [Background] Celebi N, Celebioglu B, Selcuk M, Canbay O, Karagoz AH, Aypar U. The role of antifibrinolytic agents in gynecologic cancer surgery. Saudi Med J. 2006 May;27(5):637-41. PMID 16680252
- [Background] Lundin ES, Johansson T, Zachrisson H, Leandersson U, Backman F, Falknas L, Kjolhede P. Single-dose tranexamic acid in advanced ovarian cancer surgery reduces blood loss and transfusions: double-blind placebo-controlled randomized multicenter study. Acta Obstet Gynecol Scand. 2014 Apr;93(4):335-44. doi: 10.1111/aogs.12333. Epub 2014 Feb 25. PMID 24428857
- [Background] FDA Information on Cyklokapron (tranexamic acid injection) Retrieved11/15/2015, from http://www.accessdata.fda.gov/drugsatfda_docs/label/2011/019281s030lbl.pdf